CLINICAL TRIAL: NCT00886392
Title: Distribution of Macular Edema Severity Level at the Moment of Diagnosis
Brief Title: Diabetic Macular Edema Severity at Diagnosis
Status: Completed | Type: Observational
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Virgilio Lima Gomez, Hospital Juarez de Mexico
Other Study IDs: HJM 1449/08.02.13
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Macular Edema
Keywords: Clinically Significant Macular Edema; Diabetic Macular Edema; Optical Coherence Tomography; Diabetic Retinopathy; Severity
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy; Macular Edema

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic macular edema: Type 2 diabetes patients who had clinically significant macular edema by the criterion of the ETDRS

SUMMARY:
The purpose of this study is to identify the severity level distribution at the moment of diagnosis, in diabetic patients with macular edema from a Mexico City sample, and to identify the rate with severe macular edema that needed immediate treatment.

DETAILED DESCRIPTION:
The international severity scale grades macular edema as mild, moderate or severe, according to the distance of the thickening from the center of the fovea; However, this scale does not define the distances which fulfill the criteria of "distant from" or "approaching" the center of the macula; a quantitative and reproducible tool, such as optical coherence tomography (OCT), could be more accurate to grade severity, by localizing thickening in a standardized way.

As far as we know, distribution of clinically significant macular edema at the moment of diagnosis, according to the international scale has not been described. A study was conducted to identify the rate of eyes that had severe macular edema at the moment of diagnosis, whose risk of visual loss could be higher and required immediate treatment.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic
* regardless of diabetes duration and retinopathy severity level
* one or both eyes with CSME

Exclusion Criteria:

* media opacities that prevented an adequate fast macular map from being acquired
* a thickened posterior vitreous
* any additional retinal disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population were type 2 diabetic patients with CSME who attended general hospitals of Mexico City and its metropolitan area; available population were patients with CSME evaluated at a general hospital
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Thickening measured by optical coherence tomography in 3 zones: central subfield (when field 1 was thickened), inner ring (when any of fields 2, 3, 4 or 5 was thickened), and inner ring or outer ring (when any of fields 6, 7, 8, or 9 was thickened) | at the diagnosis moment

SECONDARY OUTCOMES:
Severity level: adaptation of International clinical diabetic macular edema severity scale to fields of the OCT; mild if thickening exclusively involved outer-ring, moderate if was in inner-ring without involvement field 1, and severe if was in field 1 | at the diagnosis moment

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Muñoz Ibarra, MD, Principal Investigator — Hospital Juarez de Mexico; Dulce M Razo Blanco Hernandez, MD, Study Director — Hospital Juarez de Mexico; Virgilio Lima Gomez, MD, MsC, Study Chair — Hospital Juarez de Mexico
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico